CLINICAL TRIAL: NCT02531971
Title: Absolute Bioavailability/ Pharmacokinetic and Residual Drug Analysis of Duragesic ® Transdermal System and Generic Fentanyl Transdermal System in Healthy Adults
Brief Title: Fentanyl Patch Pharmacokinetics in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HP-00063835
Record Dates: First submitted 2015-08-19; First posted 2015-08-25 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Peer Review, Research
Keywords: Bioequivalence; Therapeutic Equivalency
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl citrate (36 h), Duragesic (192 h), Mylan (192 h) (Active Comparator): Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I) and blood samples obtained 0-36 h, washout at least one week, then wore a Duragesic® fentanyl TDDS (25 µg/h) for 72 h (Study Session II) and blood samples obtained 0-192 h, washout at least one week, then wore a Mylan fentanyl TDDS (25 µg/h) for 72 h (Study Session III) and blood samples obtained 0-192 h
  Interventions: Drug: Intravenous fentanyl citrate; Drug: Duragesic®; Drug: Mylan generic fentanyl
- Fentanyl citrate (36 h), Mylan (192 h), Duragesic (192 h) (Active Comparator): Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I) and blood samples obtained 0-36 h, washout at least one week, then wore a Mylan fentanyl TDDS (25 µg/h) for 72 h (Study Session II) and blood samples obtained 0-192 h, washout at least one week, then wore a Duragesic® fentanyl TDDS (25 µg/h) for 72 h (Study Session III) and blood samples obtained for 0-192 h
  Interventions: Drug: Intravenous fentanyl citrate; Drug: Duragesic®; Drug: Mylan generic fentanyl

INTERVENTIONS:
Drug: Intravenous fentanyl citrate — 100 micrograms (2 millilitres) via intravenous injection
Drug: Duragesic® — TDDS dosage is 25 micrograms/hour (worn for 72 h)
  Other Names: Duragesic® fentanyl skin patch
Drug: Mylan generic fentanyl — TDDS dosage is 25 micrograms/hour (worn for 72 h)
  Other Names: Mylan generic fentanyl skin patch

SUMMARY:
The study to be performed will utilize already FDA-approved marketed products in healthy adults for the purpose to generate data for establishing rate of drug delivery comparisons between RLD (reference listed drug) Duragesic ® TDDS (transdermal drug delivery system) and Generic Fentanyl TDDS in healthy adults and to ensure safety of individuals utilizing these types of products.

DETAILED DESCRIPTION:
Transdermal drug delivery systems (TDDS) available in the form of patches are convenient, attractive, and easy to use systems. Fentanyl patches are very popular TDDS available on the United States market today. Accurate determination of the rate and extent of drug release and absorption is crucial to ensure the safety of individuals using these and other types of patches. Delivery rate can be determined early in the development process by using in vitro skin flux permeation studies, and later in humans by accurately quantifying residual drug from patches post-wear and in pharmacokinetic studies. In this proposal, we will employ two types of evaluation to determine the rate and extent of drug release and absorption from RLD (reference listed drug) Duragesic ® TDDS (transdermal drug delivery system) and Generic Fentanyl TDDS, namely residual drug analysis post-wear and pharmacokinetic analysis in healthy adult volunteers. In addition, we will compare the plasma drug concentrations following patch and intravenous administration of Fentanyl, in order to determine the absolute bioavailability of these patches. We will conduct residual drug analysis of TDDS following in vivo wear using highly sensitive validated quantification methods. Positive outcome of this project will identify appropriate methods to determine the rate and extent of drug release and absorption from TDDS, and will help regulatory agencies in the development of Guidances for Industry regarding the characterization of drug release and absorption kinetics to ensure the safety of individuals utilizing these types of products

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women of any ethnic background between the age of 18 and 45 years old
2. Subjects must be non-smokers (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g. cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes) over the previous 2 months and are not currently using tobacco products
3. Provide written informed consent before initiation of any study procedures
4. Available for follow-up for the planned duration of the study
5. Able to communicate well with the investigators
6. Able to adhere to the study protocol schedule, study restrictions and examination schedule
7. Subjects who are within their ideal body weight (BMI between >17 and ≤28 kg/m2)
8. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination and medication history
9. Subjects have no history of the following: ongoing acute or intermittent pain, postoperative pain, respiratory compromise, acute or severe asthma, or constipation (less than 1 bowel movement every 2 days)
10. Negative urine drug screening test at the time of screening
11. Have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, ALT (liver function), AST (liver function) and bilirubin
12. Have normal screening laboratories for urine protein and urine glucose
13. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year [no bleeding for 12 consecutive months], or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of the first day of each study session, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or a vasectomized parter
14. Agrees not to participate in another clinical study/trial during the study period or to participate in an investigational drug study for at least one month after last study session
15. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 3 months after last study day
16. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute)
17. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-140 mmHg
    * Diastolic blood pressure 60-90 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-18 breaths per minute

Exclusion Criteria:

1. Women who are pregnant, lactating or breast feeding or have a positive serum pregnancy test at enrollment or positive urine pregnancy test on the morning of the first day of any study session
2. Smokers (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g. cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes)
3. Participation in any ongoing investigational drug trial/study or clinical drug trial/study
4. History of chronic obstructive pulmonary disease or cor pulmonale, or substantially decreased respiratory reserve, hypoxia, hypercapnia or pre-existing respiratory depression
5. Active positive Hepatitis B, C and HIV serologies
6. Positive urine drug screening test
7. Use of any prescription medication during the session 0 to 30 days or over-the counter medication e.g. antihistamines or topical corticosteroids (vitamin, herbal supplements and birth control medications not included) during the session 0 to 3 days before entry to the study
8. Use of medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product or agents deemed to be immunosuppressive as determined by physician investigator with 72 hours prior to dosing (e.g. antihistamines, systemic or topical corticosteroids (within 3 weeks prior to dosing), cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin (BCG), monoclonal antibodies, radiation therapy)
9. Use of monoamine oxidase inhibitors 21 days prior to study
10. Current use of mixed agonist/antagonist (such as pentazocine, nalbuphine or butorphanol) and partial agonist (buprenorphine) analgesics
11. Current use of anticholinergics or other medications with anticholinergic activity
12. Consumption of beverages containing alcohol, grapefruit juice, Seville oranges, or quinine (e.g. tonic water) or foods containing poppy seeds in the last 72 hours.
13. Donation or loss of greater than one pint of blood within 60 days of entry to the study
14. Any prior serious adverse reaction or hypersensitivity to fentanyl, morphine, codeine, hydrocodone, hydromorphone, oxycodone, oxymorphone, naltrexone or naloxone or any of the inactive ingredients in the TDDS (polyester/ethyl vinyl acetate, polyacrylate adhesive, silicone adhesive, dimethicone NF, or polyolefin)
15. Have a diagnosis of schizophrenia or other major psychiatric diagnosis or mental illness (e.g. major depression)
16. Medical history of personal drug or alcohol addiction or abuse
17. Any condition that would, in the opinion of the MAI, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
18. Inability to communicate or cooperate with the investigators
19. Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application site (upper arm), sunburn, raised moles and scars, open sore, scar tissue, tattoo, or coloration that would interfere with placement of test articles, skin assessment, or reactions to drug
20. Failure to pass opioid dependence challenge test on the first day study day of any study session (i.e., before taking the first dose of naltrexone hydrochloride). Each subject will be injected subcutaneously with naloxone hydrochloride (0.8 mg injection) and will be observed for 45 minutes for signs and symptoms of opioid withdrawal.
21. Within 4 weeks prior to dosing, use of medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product or agents deemed to be immunosuppressive as determined by physician investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra Stinchcomb, PhD, Principal Investigator — University of Maryland, School of Pharmacy; Hazem Hassan, PhD, Principal Investigator — Univerisity of Maryland, School of Pharmacy
Locations (1):
- General Clinical Research Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl Citrate (36 h), Duragesic® (192 h), Mylan (192 h): Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I) and blood samples were obtained for 0-36 h, washout at least one week, then same volunteers wore a Duragesic® fentanyl TDDS (25 µg/h) for 72 h (Study Session II) and blood samples were obtained for 0-192 h, washout at least one week, then same volunteers wore a Mylan fentanyl TDDS (25 µg/h) for 72 h (Study Session IIII) and blood samples obtained for 0-192 h
- Fentanyl Citrate (36 h), Mylan (192 h), Duragesic® (192 h): Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I) and blood samples obtained for 0-36 h, washout at least one week, then same volunteers wore a Mylan fentanyl TDDS (25 µg/h) for 72 h (Study Session II) and blood samples obtained for 0-192 h, washout at least one week, then same volunteers wore a Duragesic® fentanyl TDDS (25 µg/h) for 72 h (Study Session IIII) and blood samples were obtained for 0-192 h
Period: Overall Study
Arm/Group | Fentanyl Citrate (36 h), Duragesic® (192 h), Mylan (192 h) | Fentanyl Citrate (36 h), Mylan (192 h), Duragesic® (192 h)
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl Citrate, Then Duragesic®, Then Mylan: Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I), washout at least one week, then wore a Duragesic® fentanyl TDDS (25 µg/h) for 3 days (Study Session II), washout at least one week, then wore a Mylan fentanyl TDDS (25 µg/h) for 3 days (Study Session III)
- Fentanyl Citrate, Then Mylan, Then Duragesic®: Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I), washout at least one week, then wore a Mylan fentanyl TDDS (25 µg/h) for 3 days (Study Session II), washout at least one week, then wore a Duragesic® fentanyl TDDS (25 µg/h) for 3 days (Study Session III)
- Total: Total of all reporting groups
Arm/Group | Fentanyl Citrate, Then Duragesic®, Then Mylan | Fentanyl Citrate, Then Mylan, Then Duragesic® | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 6 | 10 | 16
  Caucasian | 1 | 1 | 2
  Asian | 3 | 1 | 4
  More than one race | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC 0-∞ ) ng∙h/mL
Description: drug concentration in serum vs. time; reflects the actual body exposure to drug after administration of a dose of the drug
Time Frame: 10 procedure days for Duragesic and Mylan arms each
Population: Reported values are for all 24 volunteers.
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Groups:
- Duragesic: Volunteers wore a Duragesic® fentanyl TDDS (25 µg/h) for 3 days (either Study Session II or Study Session III)
- Mylan: Volunteers wore a Mylan fentanyl TDDS (25 µg/h) for 3 days (Study Session II or Study Session III)
Arm/Group | Duragesic | Mylan
Number analyzed (Participants) | 24 | 24
ng∙h/mL | 60.1 (31.6) | 64.2 (35.1)

ADVERSE EVENTS:
Time Frame: 25 days (study duration); any adverse events were followed up until resolved
Description: All adverse events were category 3 (other, not serious); all were expected adverse events according to package inserts
Groups:
- Fentanyl Citrate: Volunteers received a single-dose of 100 µg fentanyl citrate infusion (Study Session I); blood samples obtained from 0-36 h
- Duragesic®: Volunteers wore a Duragesic® fentanyl TDDS (25 µg/h) for 72 h (either Study Session II or Study Session III); blood samples obtained from 0-192 h
- Mylan Generic Fentanyl: Volunteers wore a Mylan fentanyl TDDS (25 µg/h) for 72 h (either Study Session II or Study Session III); blood samples obtained from 0-192 h
Arm/Group | Fentanyl Citrate | Duragesic® | Mylan Generic Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 24/24 | 24/24 | 24/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl Citrate (N=24) | Duragesic® (N=24) | Mylan Generic Fentanyl (N=24)
Nausea (Product Issues) | 4 (4) | 2 (2) | 2 (2)
Decreased heart rate (Product Issues) | 10 (20) | 13 (53) | 13 (49)
Increased heart rate (Product Issues) | 2 (2) | 0 (0) | 4 (4)
Increased blood pressure (Product Issues) | 5 (6) | 6 (22) | 5 (10)
Decreased blood pressure (Product Issues) | 1 (2) | 6 (21) | 8 (21)
Headache (Product Issues) | 4 (4) | 5 (7) | 2 (3)
Decreased respiratory rate (Product Issues) | 6 (6) | 3 (7) | 3 (3)
Increased respiratory rate (Product Issues) | 15 (27) | 18 (39) | 11 (31)
Abdominal cramping (Product Issues) | 0 (0) | 0 (0) | 2 (2)
Pain, swelling, bruising, abrasions, erythema at IV catheter site (Investigations) | 0 (0) | 3 (3) | 3 (3)
Erythema (Product Issues) | 1 (1) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT02531971/Prot_SAP_000.pdf